CLINICAL TRIAL: NCT03050216
Title: QUILT-3.033: Haploidentical Donor Natural Killer (NK) Cell Infusion With Subcutaneous ALT-803 in Adults With Refractory or Relapsed Acute Myelogenous Leukemia
Brief Title: QUILT-3.033: Haplo NK With SQ ALT-803 for Adults With Relapsed or Refractory AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS056; MT2016-05 (Other: Masonic Cancer Center, University of Minnesota)
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Results first posted 2020-11-27 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cy, FLU, Haplo NK and ALT-803 (Experimental): Preparative Regimen of Fludarabine and Cyclophosphamide
  ALT-803 Activation of Donor NK Cells
  ALT-803 to Facilitate NK Cell Survival and Expansion
  Interventions: Biological: ALT-803

INTERVENTIONS:
Biological: ALT-803 — Preparative Regimen:
  Fludarabine 25 mg/m2 x 5 days start day -6 Cyclophosphamide 60 mg/kg x 2 days on day -5 and -4
  ALT-803 Stimulated Donor NK Cells:
  The apheresis product (collected day -1) will be enriched for NK cells with the large-scale CliniMacs® device (Miltenyi) by depletion of CD3+ cells to remove T-lymphocytes and depletion of CD19+ cells to remove B-lymphocytes. The NK cell enriched product will be stimulated by overnight incubation with 36.1 ng/mL ALT-803 under GMP conditions and infused on day 0.
  ALT-803 to Facilitate NK Cell Survival and Expansion:
  ALT-803 at 10 mcg/kg subcutaneously (SC) with the 1st dose administered on day 0 (no sooner than 4 hours post NK cells), day +5 and day +10 for 3 doses total

SUMMARY:
This is a multi-institutional Simon's optimal two-stage phase II trial of CD3/CD19 depleted, ALT-803 activated, haploidentical donor NK cells and subcutaneous ALT-803 given after lymphodepleting chemotherapy (CY/FLU) for the treatment of refractory or released acute myelogenous leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) and meets one of the following disease criteria:

  * Primary induction failure:

    * De novo AML - no CR after 2 or more chemotherapy induction attempts
    * Secondary AML (from MDS or treatment related): no CR after 1 or more chemotherapy induction attempts
  * Relapse after chemotherapy: not in CR after 1, 2, or 3 re-induction attempts

    * Patients > 60 years of age, the 1 cycle of chemotherapy is not required
  * Relapse after hematopoietic stem cell transplant:

    * Relapse must have occurred > 18 months after transplant
    * No re-induction required and no more than 1 re-induction attempt is allowed
* Notes:

  1. For hypomethylating agents (i.e. decitabine, azacitidine) to count as an induction/re-induction attempt, the patient must have completed a minimum of 3 monthly cycles
  2. For targeting agents (i.e. sorafenib) to count as an induction/re-induction attempt, the patient must have completed a minimum of 1 month without attaining CR
  3. 7+3 followed by 5+2 counts as TWO induction attempts
  4. Use of hydroxyurea is permitted to control blasts until Day -3 per Section 8.7
  5. A history of AML related CNS involvement is allowed if CSF analysis is negative on 2 test dates at least 2 weeks apart prior to study treatment. The use of ongoing CNS maintenance therapy is allowed while on study.
* HLA-haploidentical related donor (aged 12 to 75 years) with donor/recipient match based on a minimum of intermediate resolution DNA based Class I typing of the A and B locus (at least 2/4 class I allele)
* Karnofsky Performance Status ≥ 60%
* Adequate organ function within 14 days of study registration (28 days for pulmonary and cardiac) defined as:

  * Creatinine: ≤ 2.0 mg/dL
  * Hepatic: AST and ALT < 3 x upper limit of institutional normal
  * Pulmonary Function: oxygen saturation ≥ 90% on room air; PFT's required only if symptomatic or prior known impairment - must have pulmonary function >50% corrected DLCO and FEV1.
  * Cardiac Function: LVEF ≥ 40% by echocardiography, MUGA or cardiac MRI, no uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Able to be off prednisone or other systemic immunosuppressive medications for at least 3 days prior to NK cell infusion (excluding preparative regimen pre-medications) .
* Sexually active females of child bearing potential and males with partners of child bearing potential must agree to use effective contraception during therapy and for 4 months after completion of therapy .
* Voluntary written consent prior to the performance of any research related procedures.

Exclusion Criteria:

* Acute leukemias of ambiguous lineage
* Pregnant or breastfeeding - The agents used in this study include those that fall under Pregnancy Category D - have known teratogenic potential. Women of child bearing potential must have a negative pregnancy test at screening
* Active autoimmune disease requiring systemic immunosuppressive therapy
* History of severe asthma and currently on systemic chronic medications (mild asthma requiring inhaled steroids only is eligible)
* New or progressive pulmonary infiltrates on screening chest X-ray or chest CT scan unless cleared for study by Pulmonary. Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections).
* Uncontrolled bacterial, fungal or viral infections including HIV-1/2 or active hepatitis C/B - chronic asymptomatic viral hepatitis is allowed
* Received any investigational agent within the 14 days before the start of study treatment (1st dose of fludarabine)
* Prior ALT-803

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Berrien-Elliott MM, Becker-Hapak M, Cashen AF, Jacobs M, Wong P, Foster M, McClain E, Desai S, Pence P, Cooley S, Brunstein C, Gao F, Abboud CN, Uy GL, Westervelt P, Jacoby MA, Pusic I, Stockerl-Goldstein KE, Schroeder MA, DiPersio JF, Soon-Shiong P, Miller JS, Fehniger TA. Systemic IL-15 promotes allogeneic cell rejection in patients treated with natural killer cell adoptive therapy. Blood. 2022 Feb 24;139(8):1177-1183. doi: 10.1182/blood.2021011532. PMID 34797911

RESULTS

PARTICIPANT FLOW:
Groups:
- Cy, FLU, Haplo NK and ALT-803: Fludarabine 25 mg/m2 x 5 days start Day -6 ; Cyclophosphamide 60 mg/kg x 2 days on Day -5 and -4 ; The Alt-803 stimulated NK cell enriched product on Day 0 followed by ALT-803 at 10 mcg/kg subcutaneously on Day 0, Day 5 and Day 10
Period: Overall Study
Arm/Group | Cy, FLU, Haplo NK and ALT-803
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cy, FLU, Haplo NK and ALT-803
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Remission With or Without Incomplete Platelet Recovery
Description: To estimate the rate of complete remission with incomplete platelet recovery (CRp) - defined as leukemic clearance and neutrophil recovery without platelet recovery - by day 42 after the infusion of CD3/CD19 depleted, ALT-803 stimulated, donor NK cells and subcutaneous ALT-803 given after a non-myeloablative preparative regimen for the treatment of refractory or released acute myelogenous leukemia (AML)
Time Frame: Day 42 post NK cell infusion
Population: One patient died after receiving 2 days of chemotherapy and never received any elements of research, NK cells or ALT-803. So only 7 participants' data were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Cy, FLU, Haplo NK and ALT-803
Number analyzed (Participants) | 7
Participants | 1

2. Secondary Outcome: Incidence of in Vivo Expansion ≥100 of Donor Derived NK Cells Per /μl Blood
Description: Number of patients with successful in vivo NK-cell expansion which is defined by measuring an absolute circulating donor-derived NK cell count of ≥100 cells/μl in patient's peripheral blood.
Time Frame: Day 14 post NK cell infusion
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cy, FLU, Haplo NK and ALT-803
Number analyzed (Participants) | 7
Participants | 0

3. Secondary Outcome: Number of Participants Experiencing ALT-803 Associated Toxicity
Description: Toxicity will be classified and graded according to NCI's Common Terminology Criteria for Adverse Events V 4.0 (CTCAE)
Time Frame: Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cy, FLU, Haplo NK and ALT-803
Number analyzed (Participants) | 7
Participants | 2

4. Secondary Outcome: Number of Participants Experiencing ALT-803 Associated Toxicity
Description: Toxicity will be classified and graded according to NCI's Common Terminology Criteria for Adverse Events V 4.0 (CTCAE)
Time Frame: Day 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cy, FLU, Haplo NK and ALT-803
Number analyzed (Participants) | 7
Participants | 1

5. Secondary Outcome: Number of Participants Experiencing ALT-803 Associated Toxicity
Description: Toxicity will be classified and graded according to NCI's Common Terminology Criteria for Adverse Events V 4.0 (CTCAE)
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cy, FLU, Haplo NK and ALT-803
Number analyzed (Participants) | 7
Participants | 3

6. Secondary Outcome: Number of Participants Experiencing ALT-803 Associated Toxicity
Description: Toxicity will be classified and graded according to NCI's Common Terminology Criteria for Adverse Events V 4.0 (CTCAE)
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cy, FLU, Haplo NK and ALT-803
Number analyzed (Participants) | 7
Participants | 3

7. Secondary Outcome: Number of Participants With Treatment Related Mortality
Description: To evaluate the safety of the therapy as measured by rate of treatment related mortality (TRM) at 6 months
Time Frame: 6 months post-therapy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cy, FLU, Haplo NK and ALT-803
Number analyzed (Participants) | 7
Participants | 6

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cy, FLU, Haplo NK and ALT-803
All-Cause Mortality (participants affected / at risk) | 8/8
Serious Adverse Events (participants affected / at risk) | 7/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cy, FLU, Haplo NK and ALT-803 (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia - Changed to levaquin and micafungin (Blood and lymphatic system disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cy, FLU, Haplo NK and ALT-803 (N=8)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (6)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 7 (11)
Fatigue (General disorders) | 4 (7)
Fever (General disorders) | 5 (17)
Injection site reaction (General disorders) | 7 (24)
Pain (General disorders) | 2 (4)
Infusion related reaction (General disorders) | 3 (3)
Clostridium Difficile Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (3)
Urine output decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 6 (12)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) — lightheadedness
Anxiety (Psychiatric disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2) — Diffuse lace type rash with associated itching
Hypertension (Vascular disorders) | 4 (14)
Hypotension (Vascular disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT03050216/Prot_SAP_000.pdf